CLINICAL TRIAL: NCT00718016
Title: Assessment of the Cyberlink Control System for Use by the ALS Patient
Brief Title: Assessment of the Cyberlink Control System for Use by the Amyotrophic Lateral Sclerosis (ALS) Patient
Status: Terminated | Type: Observational
Why Stopped: New protocol was developed based on preliminary results from this study.
Sponsor: Drexel University College of Medicine (Other)
Collaborators: MDA/ALS Center of Hope (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Other Study IDs: Internal-903
Record Dates: First submitted 2008-07-14; First posted 2008-07-18 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Neurodegenerative Disease; Motor Neuron Disease
Keywords: Amyotrophic Lateral Sclerosis; Cerebrospinal Fluid; Neurodegenerative Disease; Motor Neuron Disease; Autonomic Nervous System; Neurodegenerative Diseases; Movement Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Motor Neuron Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALS: Subjects having either definite or probable ALS by El Escorial Criteria.

SUMMARY:
The goal of this project is to determine whether this device is a practical and realistic means for ALS patients to operate their computers with only the use of facial, brainwave, and eye movements. This study is intended to evaluate both the complexity of the system and the degree to which complications of ALS (such as severity of involuntary movements) may interfere with the use of cyberlink.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 18-75 diagnosed with probable or definite ALS.

Exclusion Criteria:

* Those with decision impairment will not be considered.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALS clinic patients at MDA/ALS Center of Hope.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2004-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Usability of the Cyberlink System | 4 1-hr sessions
  Reliability and accuracy of the Cyberlink System at the end of the 4th session will be used to assess overall usability of the system

CONTACTS AND LOCATIONS:
Overall Officials: Terry Heiman-Patterson, MD, Study Director — MDA/ALS Center of Hope
Locations (1):
- MDA/ALS Center of Hope, Philadelphia, Pennsylvania, United States